CLINICAL TRIAL: NCT00763711
Title: Injectable Bulking Agent Needle Guide
Acronym: NG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Carbon Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1006
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Urinary Incontinence; Intrinsic Sphincter Deficiency
Keywords: Urinary Incontinence; ISD
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injection with Needle Guide (Experimental)
  Interventions: Device: Needle Guided Periurethral Injection

INTERVENTIONS:
Device: Needle Guided Periurethral Injection — Bulking Agent injection using a needle guide

SUMMARY:
The purpose of this study is to evaluate the use of the Needle Guide as an assist in properly guiding an injection needle into the appropriate tissue plane during an injectable bulking agent procedure in women using a FDA approved injectable bulking agent. The injectable bulking agent will be Durasphere EXP.

ELIGIBILITY:
Individuals satisfying the "Indications" and "Contraindications" criteria in the Durasphere EXP Directions for Use may participate.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
to evaluate the consistency of the location of the injection site and resulting location of bulking effect | at procedure
Safety will be demonstrated through an analysis of morbidity and complication rates, (if any), associated with the use of the Needle Guide. | 1 week

SECONDARY OUTCOMES:
to evaluate the comparative ease of the injection procedure using the Bulking Agent Needle Guide as compared to the traditional transurethral or periurethral injection technique. | at procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dean Klein, Study Director — Carbon Medical Technologies
Locations (2):
- United States (2):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Advanced Urogynecology, West Chester, Ohio

REFERENCES:
- See also: Related Info — http://carbonmed.com